CLINICAL TRIAL: NCT02438371
Title: Nifedipine Alone or Nifedipine Plus Indomethacin for Treatment of Acute Preterm Labor: An Open Label, Randomized Comparative Effectiveness Controlled Trial
Brief Title: Nifedipine or Nifedipine Plus Indomethacin for Treatment of Acute Preterm Labor
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study halted due to slow recruitment
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Jerrie Refuerzo, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-15-0134
Record Dates: First submitted 2015-05-05; First posted 2015-05-08 (Estimated); Results first posted 2021-11-24 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-10

CONDITIONS: Preterm Labor
Keywords: pregnancy; preterm labor; tocolysis
MeSH Terms: conditions — Obstetric Labor, Premature | interventions — Nifedipine; Indomethacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nifedipine (Active Comparator): Participants will receive nifedipine 10 mg orally every 20 minutes for 3 doses, then nifedipine 10 mg every 6 hours for a total of 48 hours.
  Interventions: Drug: Nifedipine
- Nifedipine plus Indomethacin (Active Comparator): Participants will receive will receive nifedipine 10 mg orally every 20 minutes for 3 doses, then nifedipine 10 mg every 6 hours for a total of 48 hours, as well as indomethacin 100 mg orally, then indomethacin 50 mg orally every 6 hours for a total of 48 hours.
  Interventions: Drug: Nifedipine; Drug: Indomethacin

INTERVENTIONS:
Drug: Nifedipine
  Other Names: Procardia
Drug: Indomethacin
  Arms: Nifedipine plus Indomethacin

SUMMARY:
Tocolytic agents are used for the treatment of preterm labor. It is unclear whether combination treatments of two tocolytic agents are more effective in stopping preterm labor compared to one. Therefore, the investigators propose a comparative effective trial of nifedipine plus indomethacin vs. nifedipine alone for the treatment of preterm labor

DETAILED DESCRIPTION:
The investigators current treatment for preterm labor has not been shown to be effective in prolonging pregnancy sufficiently to improve neonatal outcomes and other treatment strategies are needed. Multiple examples demonstrate that multi-agent treatments are routine clinical practice in other fields of medicine including chemotherapeutics for cancer, multi-therapeutics for myocardial infarction and broad spectrum antibiotics for pneumonia. At this time, it is unclear if a combination of tocolytic medications for preterm labor is more advantageous for women. If pregnancy is prolonged with combined tocolytic therapy, this could directly influence the treatment of preterm labor and potentially improve neonatal outcomes. There currently are no trials of combination regimens using widely used tocolytic agents, such as nifedipine and indomethacin. Thus, we propose a comparative effective trial of nifedipine plus indomethacin vs. nifedipine alone for the treatment of preterm labor

ELIGIBILITY:
Inclusion Criteria:

* We will include pregnant women between 22 0/7 to 31 6/7 weeks gestation who present with regular uterine contractions defined as at least one contraction every 10 minutes for 30 minutes with at least one of the following:
* cervical change of at least 1 cm or
* cervical dilation of 2 cm at the time of initial exam or
* positive fetal fibronectin and transvaginal cervical length <2.5 cm

Exclusion Criteria:

* We will exclude pregnant women with any contraindication to tocolysis:
* clinical chorioamnionitis (defined as a temperature of >100.4 F and any of the following: fundal tenderness, maternal tachycardia, fetal tachycardia or purulent vaginal discharge)
* non reassuring fetal heart tones
* suspected placental abruption
* preterm premature rupture of membranes
* prior tocolytic treatment during the past 48 hours
* known adverse effect to indomethacin or nifedipine
* already receiving nifedipine for chronic hypertension

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2019-10-10 (Actual); Study Completion 2019-10-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Hutchinson, M.S., Study Director — The University of Texas Health Science Center, Houston
Locations (1):
- Memorial Hermann Hospital Texas Medical Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wilson A, Hodgetts-Morton VA, Marson EJ, Markland AD, Larkai E, Papadopoulou A, Coomarasamy A, Tobias A, Chou D, Oladapo OT, Price MJ, Morris K, Gallos ID. Tocolytics for delaying preterm birth: a network meta-analysis (0924). Cochrane Database Syst Rev. 2022 Aug 10;8(8):CD014978. doi: 10.1002/14651858.CD014978.pub2. PMID 35947046

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The numbers listed in the Participant Flow section correspond to maternal participants.
Groups:
- Nifedipine: Participants will receive nifedipine 10 mg orally every 20 minutes for 3 doses, then nifedipine 10 mg every 6 hours, for a total of 48 hours.
- Nifedipine Plus Indomethacin: Participants will receive will receive nifedipine 10 mg orally every 20 minutes for 3 doses, then nifedipine 10 mg every 6 hours, for a total of 48 hours, as well as indomethacin 100 mg orally, then indomethacin 50 mg orally every 6 hours, for a total of 48 hours.
Period: Overall Study
Arm/Group | Nifedipine | Nifedipine Plus Indomethacin
Started | 24 | 25
Received Intervention | 24 | 25
Completed | 20 | 22
Not Completed | 4 | 3
Not completed — Lost to Follow-up | 3 | 2
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are reported for all who completed the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Nifedipine | Nifedipine Plus Indomethacin | Total
Number analyzed (Participants) | 20 | 22 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.0 (7.5) | 28.5 (7.7) | 28.3 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 22 | 42
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African/African American/Black American | 9 | 15 | 24
  Asian | 1 | 0 | 1
  Hispanic | 7 | 6 | 13
  White | 3 | 1 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20 | 22 | 42

OUTCOME MEASURES:

1. Primary Outcome: Number of Maternal Participants Who Achieve 48 Hours of Pregnancy Prolongation
Time Frame: 48 hours after administration of tocolytic agent
Population: Data for this outcome measure were not collected for 4 in the Nifedipine arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Nifedipine | Nifedipine Plus Indomethacin
Number analyzed (Participants) | 16 | 22
Participants | 15 | 20

2. Secondary Outcome: Number of Maternal Participants Who Achieve 7 Days of Pregnancy Prolongation
Time Frame: 7 days after administration of tocolytic agent
Population: Data for this outcome measure were not collected for 4 in the Nifedipine arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Nifedipine | Nifedipine Plus Indomethacin
Number analyzed (Participants) | 16 | 22
Participants | 12 | 18

3. Secondary Outcome: Number of Days From First Dose of Tocolytic Agent to Delivery
Description: Length of time from tocolytic initiation to the time of delivery
Time Frame: from time of tocolytic initiation to the time of delivery (from about 1 day to about 2 months)
Population: Data for this outcome measure were not collected for 4 in the Nifedipine arm.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Nifedipine | Nifedipine Plus Indomethacin
Number analyzed (Participants) | 16 | 22
days | 24.8 [6.9 to 49.8] | 42.6 [24.1 to 61.8]

4. Secondary Outcome: Neonatal Birthweight
Time Frame: at the time of birth
Population: Data for this outcome measure were not collected for 4 neonates in the Nifedipine arm and 1 neonate in the Nifedipine plus Indomethacin arm. (There are more neonates than maternal participants because 6 mothers in the Nifedipine arm had twins and 1 mother in the Nifedipine plus Indomethacin arm had twins.)
Measure: Median (Inter-Quartile Range); unit: grams
Arm/Group | Nifedipine | Nifedipine Plus Indomethacin
Number analyzed (Participants) | 22 | 22
grams | 1870.0 [1451.2 to 2317.5] | 2571.0 [1733.8 to 3073.8]

5. Secondary Outcome: Neonatal Sex
Time Frame: at the time of birth
Population: Data for this outcome measure were not collected for 4 neonates in the Nifedipine arm. (There are more neonates than maternal participants because 6 mothers in the Nifedipine arm had twins and 1 mother in the Nifedipine plus Indomethacin arm had twins.)
Measure: Count of Participants; unit: Participants
Arm/Group | Nifedipine | Nifedipine Plus Indomethacin
Number analyzed (Participants) | 22 | 23
Participants
  Female | 6 | 9
  Male | 16 | 14

6. Secondary Outcome: Number of Neonates Who Were Admitted to the Neonatal Intensive Care Unit (NICU)
Time Frame: from birth until hospital discharge or day 120 of life (whichever occurs first)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Nifedipine | Nifedipine Plus Indomethacin
Number analyzed (Participants) | 22 | 22
Participants | 16 | 13

7. Secondary Outcome: Neonatal Length of Stay in NICU
Time Frame: from birth until hospital discharge or day 120 of life (whichever occurs first)
Population: Data for this outcome measure were not collected for 10 neonates in the Nifedipine arm and 10 neonates in the Nifedipine plus Indomethacin arm. (There are more neonates than maternal participants because 6 mothers in the Nifedipine arm had twins and 1 mother in the Nifedipine plus Indomethacin arm had twins.)
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Nifedipine | Nifedipine Plus Indomethacin
Number analyzed (Participants) | 16 | 13
days | 36.3 [26.0 to 46.2] | 25.3 [14.0 to 52.2]

8. Secondary Outcome: Neonatal Length of Hospital Stay
Time Frame: from birth until hospital discharge or day 120 of life (whichever occurs first)
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Nifedipine | Nifedipine Plus Indomethacin
Number analyzed (Participants) | 22 | 22
days | 31.8 [3.0 to 44.7] | 10.9 [2.5 to 27.4]

9. Secondary Outcome: Number of Neonatal Deaths
Time Frame: from birth until hospital discharge or day 120 of life (whichever occurs first)
Population: Data for this outcome measure were not collected for 4 neonates in the Nifedipine arm and 2 neonates in the Nifedipine plus Indomethacin arm. (There are more neonates than maternal participants because 6 mothers in the Nifedipine arm had twins and 1 mother in the Nifedipine plus Indomethacin arm had twins.)
Measure: Count of Participants; unit: Participants
Arm/Group | Nifedipine | Nifedipine Plus Indomethacin
Number analyzed (Participants) | 22 | 21
Participants | 1 | 1

10. Secondary Outcome: Number of Neonates With Intraventricular Hemorrhage Diagnosed Using Cranial Ultrasonography
Time Frame: from birth until hospital discharge or day 120 of life (whichever occurs first)
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Nifedipine | Nifedipine Plus Indomethacin
Number analyzed (Participants) | 22 | 21
Participants | 3 | 2

11. Secondary Outcome: Number of Neonates With Necrotizing Enterocolitis
Time Frame: from birth until hospital discharge or day 120 of life (whichever occurs first)
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Nifedipine | Nifedipine Plus Indomethacin
Number analyzed (Participants) | 22 | 21
Participants | 2 | 0

12. Secondary Outcome: Number of Neonates With Culture-positive Sepsis
Time Frame: from birth until hospital discharge or day 120 of life (whichever occurs first)
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Nifedipine | Nifedipine Plus Indomethacin
Number analyzed (Participants) | 22 | 21
Participants | 3 | 3

13. Secondary Outcome: Number of Neonates With Seizures
Time Frame: from birth until hospital discharge or day 120 of life (whichever occurs first)
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Nifedipine | Nifedipine Plus Indomethacin
Number analyzed (Participants) | 22 | 21
Participants | 0 | 1

14. Secondary Outcome: Number of Neonates Who Needed Mechanical Ventilation
Time Frame: from birth until hospital discharge or day 120 of life (whichever occurs first)
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Nifedipine | Nifedipine Plus Indomethacin
Number analyzed (Participants) | 22 | 21
Participants | 4 | 3

15. Secondary Outcome: Neonatal Duration of Ventilator Use
Time Frame: from birth until hospital discharge or day 120 of life (whichever occurs first)
Population: Data for this outcome measure were not collected for 22 neonates in the Nifedipine arm and 20 neonates in the Nifedipine plus Indomethacin arm. (There are more neonates than maternal participants because 6 mothers in the Nifedipine arm had twins and 1 mother in the Nifedipine plus Indomethacin arm had twins.)
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Nifedipine | Nifedipine Plus Indomethacin
Number analyzed (Participants) | 4 | 3
hours | 32.5 [25.4 to 414.8] | 186.0 [103.0 to 1593.0]

16. Secondary Outcome: Number of Neonates Who Received Continuous Positive Airway Pressure (CPAP)
Time Frame: from birth until hospital discharge or day 120 of life (whichever occurs first)
Population: Data for this outcome measure were not collected for 5 neonates in the Nifedipine arm and 2 neonates in the Nifedipine plus Indomethacin arm. (There are more neonates than maternal participants because 6 mothers in the Nifedipine arm had twins and 1 mother in the Nifedipine plus Indomethacin arm had twins.)
Measure: Count of Participants; unit: Participants
Arm/Group | Nifedipine | Nifedipine Plus Indomethacin
Number analyzed (Participants) | 21 | 21
Participants | 11 | 8

17. Secondary Outcome: Number of Maternal Participants Who Delivered by Cesarean Delivery
Time Frame: at the the time of birth
Population: Data for this outcome measure were not collected for 4 in the Nifedipine arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Nifedipine | Nifedipine Plus Indomethacin
Number analyzed (Participants) | 16 | 22
Participants | 5 | 5

18. Secondary Outcome: Number of Maternal Participants Who Had Clinical Chorioamnionitis
Time Frame: from time of tocolytic initiation to the time of delivery (from about 1 day to about 2 months)
Population: Data for this outcome measure were not collected for 4 in the Nifedipine arm and 1 in the Nifedipine plus Indomethacin arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Nifedipine | Nifedipine Plus Indomethacin
Number analyzed (Participants) | 16 | 21
Participants | 1 | 0

19. Secondary Outcome: Number of Maternal Participants Who Had Preterm Premature Rupture of Membranes (PPROM)
Time Frame: from time of tocolytic initiation to the time of delivery (from about 1 day to about 2 months)
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | Nifedipine | Nifedipine Plus Indomethacin
Number analyzed (Participants) | 16 | 21
Participants | 2 | 2

20. Secondary Outcome: Number of Maternal Participants Who Had Preeclampsia
Time Frame: from time of tocolytic initiation to the time of delivery (from about 1 day to about 2 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Nifedipine | Nifedipine Plus Indomethacin
Number analyzed (Participants) | 20 | 22
Participants | 1 | 2

21. Secondary Outcome: Number of Maternal Participants Who Needed Blood Transfusion
Time Frame: from time of birth to time of discharge from hospital (about 2-3 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Nifedipine | Nifedipine Plus Indomethacin
Number analyzed (Participants) | 20 | 22
Participants | 1 | 1

22. Secondary Outcome: Number of Maternal Participants With Headache
Time Frame: from time of tocolytic initiation to the time of hospital discharge (from about 2 days to about 2 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Nifedipine | Nifedipine Plus Indomethacin
Number analyzed (Participants) | 20 | 22
Participants | 0 | 1

23. Secondary Outcome: Number of Maternal Participants With Nausea
Time Frame: from time of tocolytic initiation to the time of hospital discharge (from about 2 days to about 2 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Nifedipine | Nifedipine Plus Indomethacin
Number analyzed (Participants) | 20 | 22
Participants | 1 | 0

24. Secondary Outcome: Number of Maternal Participants With Vomiting
Time Frame: from time of tocolytic initiation to the time of hospital discharge (from about 2 days to about 2 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Nifedipine | Nifedipine Plus Indomethacin
Number analyzed (Participants) | 20 | 22
Participants | 0 | 0

25. Secondary Outcome: Number of Maternal Participants With Acid Reflux
Time Frame: from time of tocolytic initiation to the time of hospital discharge (from about 2 days to about 2 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Nifedipine | Nifedipine Plus Indomethacin
Number analyzed (Participants) | 20 | 22
Participants | 1 | 1

26. Secondary Outcome: Number of Maternal Participants With Hypotension
Time Frame: from time of tocolytic initiation to the time of hospital discharge (from about 2 days to about 2 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Nifedipine | Nifedipine Plus Indomethacin
Number analyzed (Participants) | 20 | 22
Participants | 1 | 1

27. Secondary Outcome: Number of Maternal Participants With Tachycardia
Time Frame: from time of tocolytic initiation to the time of hospital discharge (from about 2 days to about 2 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Nifedipine | Nifedipine Plus Indomethacin
Number analyzed (Participants) | 20 | 22
Participants | 1 | 1

28. Secondary Outcome: Number of Maternal Participants With Syncope
Time Frame: from time of tocolytic initiation to the time of hospital discharge (from about 2 days to about 2 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Nifedipine | Nifedipine Plus Indomethacin
Number analyzed (Participants) | 20 | 22
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Maternal participants: from time of tocolytic initiation to the time of hospital discharge (from about 2 days to about 2 months) Neonates: from birth until hospital discharge or day 120 of life (whichever occurs first)
Description: Adverse Events are reported for 20 maternal participants and 26 neonates in the Nifedipine arm (6 mothers in the Nifedipine arm had twins) and are reported for 22 maternal participants and 23 neonates in the Nifedipine Plus Indomethacin arm (1 mother in the Nifedipine Plus Indomethacin arm had twins). The 2 deaths were neonatal deaths (there were no maternal deaths).
Arm/Group | Nifedipine | Nifedipine Plus Indomethacin
All-Cause Mortality (participants affected / at risk) | 1/46 | 1/45
Serious Adverse Events (participants affected / at risk) | 24/46 | 38/45
Other Adverse Events (participants affected / at risk) | 4/46 | 4/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Nifedipine (N=46) | Nifedipine Plus Indomethacin (N=45)
Death (neonatal) (General disorders) | 1/26 (1) | 1/23 (1)
Admission to NICU (neonatal) (General disorders) | 16/26 (16) | 13/23 (13)
Intraventricular Hemorrhage (neonatal) (Vascular disorders) | 3/26 (3) | 2/23 (2)
Necrotizing Enterocolitis (neonatal) (Infections and infestations) | 2/26 (2) | 0/23 (0)
Culture-Positive Sepsis (neonatal) (Infections and infestations) | 3/26 (3) | 3/23 (3)
Seizures (neonatal) (Nervous system disorders) | 0/26 (0) | 1/23 (1)
Received Mechanical Ventilation (neonatal) (Respiratory, thoracic and mediastinal disorders) | 4/26 (4) | 3/23 (3)
Received Continuous Positive Airway Pressure (CPAP) (neonatal) (Respiratory, thoracic and mediastinal disorders) | 11/26 (11) | 8/23 (8)
Respiratory distress syndrome (RDS) (neonatal) (Respiratory, thoracic and mediastinal disorders) | 10/26 (10) | 5/23 (5)
Retinopathy of prematurity (neonatal) (Eye disorders) | 4/26 (4) | 1/23 (1)
Received Blood Transfusion (maternal) (General disorders) | 1/20 (1) | 1/22 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Nifedipine (N=46) | Nifedipine Plus Indomethacin (N=45)
Headache (maternal) (General disorders) | 0/20 (0) | 1/22 (1)
Nausea (maternal) (General disorders) | 1/20 (1) | 0/22 (0)
Acid Reflux (maternal) (Gastrointestinal disorders) | 1/20 (1) | 1/22 (1)
Hypotension (maternal) (Vascular disorders) | 1/20 (1) | 1/22 (1)
Tachycardia (maternal) (Cardiac disorders) | 1/20 (1) | 1/22 (1)
Clinical Chorioamnionitis (maternal) (Infections and infestations) | 1/20 (1) | 0/22 (0)
Preterm Premature Rupture of Membranes (PPROM) (maternal) (Pregnancy, puerperium and perinatal conditions) | 2/20 (2) | 2/22 (2)
Preeclampsia (maternal) (Pregnancy, puerperium and perinatal conditions) | 1/20 (1) | 2/22 (2)

LIMITATIONS AND CAVEATS:
Small sample size

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-02): https://cdn.clinicaltrials.gov/large-docs/71/NCT02438371/Prot_SAP_000.pdf